CLINICAL TRIAL: NCT00470314
Title: Therapeutic Efficacy of L-Ornithine L-Aspartate Infusion in Patients With Acute Liver Failure: A Double- Blind, Randomized, Placebo- Controlled Study
Brief Title: Therapeutic Efficacy of L-Ornithine L-Aspartate Infusion in Patients With Acute Liver Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GE-LOLA/2005
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-04

CONDITIONS: Acute Liver Failure
Keywords: Acute liver failure; Ornithine Aspartate; Ammonia; Encephalopathy
MeSH Terms: conditions — Liver Failure, Acute; Brain Diseases | interventions — ornithylaspartate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: L-Ornithine L-Aspartate

SUMMARY:
The purpose of the study is to determine whether L-Ornithine L-Aspartate infusion improves the survival of patients with acute liver failure.

DETAILED DESCRIPTION:
Acute liver failure (ALF) has a high mortality. However, those who survive recover completely without any sequel. Liver transplantation is logistically and financially difficult in most countries with the highest disease burden. It also entails a lifelong commitment to immunosuppression. We therefore need new treatment options to improve the survival of medically managed patients with ALF.

Ammonia is believed to be the major neurotoxin in ALF. There is experimental evidence of direct and indirect ammonia neurotoxicity in ALF. The brain does not have a urea cycle, and relies on glutamine synthesis in the astrocytes for removal of excess ammonia. Increased intracellular glutamine in the astrocytes leads to cellular swelling. Increased brain ammonia concentrations also result in altered expression of key astrocyte proteins including glial fibrillary acidic protein, glutamate and glycine transporters and "peripheral-type" (mitochondrial) BZD receptors. Accumulation of ammonia in brain results in a redistribution of cerebral blood flow from cortical to sub-cortical structures, and also has direct effects on neurotransmission. Increased ammonia concentration upregulates the peripheral-type benzodiazepine (PTBR) receptors in the outer membrane of astroglial mitochondria, and enhance the synthesis and release of neurosteroids, some of which are known GABA (A) receptor agonists.

There is now evidence of high blood ammonia levels in ALF , with a substantial blood-to-brain ammonia transfer.Brain-blood ammonia concentration ratios (normally of the order of 2) are increased up to 4 fold in liver failure. Higher ammonia levels have been co-related with higher mortality and complications in human clinical trials. Clemmesen et al found that ALF patients who died of cerebral herniation had higher ammonia levels as compared to the survivors. We have also previously shown that higher ammonia levels at admission predicts a poorer survival rate, and arterial ammonia levels are an independent predictor of mortality by logistic regression analysis. An arterial ammonia level of > 124 μmol/l was found to predict mortality with 78.6% sensitivity and 76.3% specificity.There is thus a strong rationale for using ammonia lowering therapies in ALF.

LOLA is a compound salt of Ornithine and Aspartate. The mechanism of its ammonia lowering action has been defined. LOLA provides critical substrates for both urea and glutamine synthesis- the key pathways of ammonia detoxification in the liver. Urea synthesis is carried out in a low affinity, high capacity system that exists largely in the periportal hepatocytes. In these cells, Ornithine serves as an activator of ornithine-carbamoyltransferase and carbamylphosphate-synthetase. In addition, Ornithine itself acts as a substrate for urea genesis. Hence LOLA can activate the periportal urea cycle. Glutamine synthesis is a high affinity, relatively low capacity system located in the perivenous hepatocytes. Ornithine is converted to α -ketoglutarate, and taken up by these perivenous hepatocytes and serves as a carbon source for glutamine synthesis. LOLA also upregulates glutamine synthesis in the skeletal muscle via glutamine synthetase (GS). Recently, in animal models an increased transport of ornithine across the blood brain barrier and an increase in the brain glutamine synthesis after LOLA treatment has been described, and suggests that LOLA may have both centrally (CNS) and peripherally mediated effects. , LOLA has been shown to reduce raised ammonia levels in experimental models of hyper-ammonemia, and in human cirrhotic patients. In patients with cirrhosis,LOLA improves psychometric performance and improves the mental status.

LOLA is therefore a promising agent for use in ALF patients. It has scientific rationale and has been found to be effective in cirrhosis. There is however only a single experimental study of LOLA in a rat model of acute liver injury. LOLA infusion could normalize the plasma ammonia and lead to a significant reduction in brain water content. We would like to study whether LOLA infusion in patients with ALF can reduce ammonia levels and improve survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute liver failure, as defined by the development of encephalopathy within 4 weeks of onset of symptoms in the absence of preexisting liver disease.

Exclusion Criteria:

* Presence of > 3 adverse prognostic factors (Age > 40 years, clinical evidence of cerebral edema, bilirubin >15mg/dL, and prothrombin time prolonged by > 25 seconds) at the initial patient evaluation.
* Suspicion of underlying cirrhosis.
* Previous treatment with LOLA or other ammonia lowering treatments before admission.
* Malarial hepatopathy, enteric hepatitis, alcoholic hepatitis, or ischemic hepatitis.
* Active alcohol use of >40 gm/week at the onset of illness.
* Renal insufficiency at admission, as defined by a urine output of <500 mL/d and /or creatinine level of > 3mg/dL.
* Inability to randomize within 24 hours of admission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-01; Study Completion 2007-05 (Estimated)

PRIMARY OUTCOMES:
Improvement in survival. | Within 30 days of disease onset

SECONDARY OUTCOMES:
Reduction in ammonia levels during and at the end of 72 hour LOLA infusion. | 72 hours
Improvement of encephalopathy by one or more grades. | 72 hours
Reduction of consciousness recovery time (CRT) among survivors. | Within 30 days of disease onset
Prolongation of time to death among non-survivors. | Within 30 days of disease onset
Prevention / reduction of cerebral edema. | 72 hours
Reduction of seizures frequency. | Within 30 days of disease onset

CONTACTS AND LOCATIONS:
Overall Officials: Subrat Kr Acharya, M.D., D.M., Study Director — All India Institute of Medical Sciences; Vikram Bhatia, M.D., D.M., Principal Investigator — All India Institute of Medical Sciences; Amit Singhal, M.D., Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, Delhi, India

REFERENCES:
- [Background] Bhatia V, Singh R, Acharya SK. Predictive value of arterial ammonia for complications and outcome in acute liver failure. Gut. 2006 Jan;55(1):98-104. doi: 10.1136/gut.2004.061754. Epub 2005 Jul 15. PMID 16024550
- [Background] Clemmesen JO, Larsen FS, Kondrup J, Hansen BA, Ott P. Cerebral herniation in patients with acute liver failure is correlated with arterial ammonia concentration. Hepatology. 1999 Mar;29(3):648-53. doi: 10.1002/hep.510290309. PMID 10051463
- [Background] Staedt U, Leweling H, Gladisch R, Kortsik C, Hagmuller E, Holm E. Effects of ornithine aspartate on plasma ammonia and plasma amino acids in patients with cirrhosis. A double-blind, randomized study using a four-fold crossover design. J Hepatol. 1993 Nov;19(3):424-30. doi: 10.1016/s0168-8278(05)80553-7. PMID 8151104
- [Background] Kircheis G, Nilius R, Held C, Berndt H, Buchner M, Gortelmeyer R, Hendricks R, Kruger B, Kuklinski B, Meister H, Otto HJ, Rink C, Rosch W, Stauch S. Therapeutic efficacy of L-ornithine-L-aspartate infusions in patients with cirrhosis and hepatic encephalopathy: results of a placebo-controlled, double-blind study. Hepatology. 1997 Jun;25(6):1351-60. doi: 10.1002/hep.510250609. PMID 9185752
- [Background] Rose C, Michalak A, Rao KV, Quack G, Kircheis G, Butterworth RF. L-ornithine-L-aspartate lowers plasma and cerebrospinal fluid ammonia and prevents brain edema in rats with acute liver failure. Hepatology. 1999 Sep;30(3):636-40. doi: 10.1002/hep.510300311. PMID 10462368
- [Derived] Acharya SK, Bhatia V, Sreenivas V, Khanal S, Panda SK. Efficacy of L-ornithine L-aspartate in acute liver failure: a double-blind, randomized, placebo-controlled study. Gastroenterology. 2009 Jun;136(7):2159-68. doi: 10.1053/j.gastro.2009.02.050. PMID 19505424
- See also: Comprehensive details of liver failure in the pediatric population — http://www.emedicine.com/PED/topic808.htm